CLINICAL TRIAL: NCT00291096
Title: High Risk Breast Clinic: Protocol for Women at Increased Risk for Developing Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Carol Fabian, MD (Other)
Responsible Party: Sponsor-Investigator, Carol Fabian, MD, Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Other Study IDs: 4601
Record Dates: First submitted 2006-02-10; First posted 2006-02-13 (Estimated); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer
Keywords: breast atypia; fine needle aspiration; high risk for breast cancer; breast epithelial hyperplasia
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — RPFNA specimens, serum, NAF
Oversight: Data Monitoring Committee: No

SUMMARY:
The overall goal of this project is to develop an integrative system of breast cancer risk assessment based on epidemiologic and biologic risk variables, as well as to develop or refine risk biomarkers which may be useful in predicting and monitoring response to prevention interventions.

DETAILED DESCRIPTION:
1. To correlate established risk biomarkers such as cytomorphology obtained from random periareolar fine needle aspiration ( RPFNA), mammographic breast density, serum bioavailable estradiol and IGF-1/IGFBP-3 with each other and with 5-10 year Gail risk estimates. Where available, and with appropriate safe guards to maintain status for breast cancer susceptibility genes may be included.
2. To determine the relative predictive value of established risk biomarkers for the development of DCIS and/or invasive cancer.
3. To evaluate potential new breast tissue-based biomarkers including Ki-67, PCNA, ER, COX-2, aromatase, methylation of key tumor suppressor genes (i.e., RAR, p16, etc), proteomic patterns in RPFNA and nipple aspirate fluid (NAF), as well as NAF hormone levels, and correlate them with other risk biomarkers listed in 1.
4. To determine the prevalence of polymorphisms of a panel of genes important in hormone and xenobiotic metabolism as well as DNA repair and correlate these polymorphisms with established risk biomarkers listed in 1, as well as with development of DCIS and invasive cancer.
5. To maintain contact with this initially identified cohort of high risk women, acquire demographic data, biologic specimens and data and follow them prospectively for the development.

ELIGIBILITY:
Inclusion Criteria:

* women with at least 2 times the normal risk of developing breast cancer
* between the ages of 30-65 (or within 10 years of youngest age at diagnosis in first degree relative)
* greater than six months from ingestion of antihormonal therapy
* greater than 1 year from pregnancy, lactation, or chemotherapy
* willing to have a mammogram within six months prior to RPFNA
* willing to discontinue NSAIDS or herbal supplements
* willing to have blood drawn

Exclusion Criteria:

* no metastatic malignancy of any kind
* no breast implants or tram flap reconstructions
* no radiation to both breasts
* no women who have a current mammogram or clinical breast exam suspicious for cancer

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Self-identified women at high risk for development of breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 1989-08 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Prediction of risk for developing breast cancer | ongoing
  development of algorithm for predicting risk for developing breast cancer based on random sampling of benign breast tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Carol J Fabian, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No